CLINICAL TRIAL: NCT03458962
Title: Ending the Diagnostic Odyssey: Whole Genome Sequencing (WGS) to Identify Genetic Determinants of Previously Undiagnosed Disease in Children
Brief Title: Diagnostic Odyssey: Whole Genome Sequencing (WGS)
Status: Recruiting | Type: Observational
Sponsor: Nicklaus Children's Hospital f/k/a Miami Children's Hospital (Other)
Collaborators: Rady Pediatric Genomics & Systems Medicine Institute (Other)
Responsible Party: Sponsor
Other Study IDs: (WGS) Protocol #20172859
Record Dates: First submitted 2018-03-02; First posted 2018-03-08 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-11

CONDITIONS: Genetic Disease; Genetic Syndrome
Keywords: Nicklaus Children's; Pediatric; Genomic; Precision Medicine; Biorepository; Rady Children's
MeSH Terms: conditions — Genetic Diseases, Inborn

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, saliva, tissue, left-over samples from residual blood, CSF, bone, stool, urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Genetic Enrollees: Enrollment of patients for whom WGS may be beneficial. Patients who are ill and for whom a genetic diagnosis is suspected but not yet established.
  Interventions: Genetic: Genetic Enrollees

INTERVENTIONS:
Genetic: Genetic Enrollees — Identification of new genetic diagnoses in children with multiple congenital anomalies, developmental delay, autism, seizures, intellectual disabilities, neurodegenerative disorders and metabolic illness. Samples and data will be stored in a pediatric biorepository. A subset of samples will undergo genetic/genomic analysis.

SUMMARY:
The goal of this collaborative research is to study human genomes in children with suspected congenital disease, multiple-congenital anomalies and/or multi-organ disease of unknown etiology by understanding the potential value of Whole Genome Sequencing (WGS) in establishing genetic diagnosis. The study will examine diagnosis rates, changes in clinical care as a result of a genetic diagnosis, health economics including potential cost-effectiveness of WGS and patient and provider experience with genomic medicine.

DETAILED DESCRIPTION:
The goal of this collaborative research is to study human genomes in children with suspected congenital disease, multiple-congenital anomalies and/or multi-organ disease of unknown etiology, in order to understand the potential value of WGS in establishing a genetic diagnosis. The study will examine diagnosis rates, changes in clinical care as a result of a genetic diagnosis, health economics including potential cost-effectiveness of WGS, and patient and provider experience with genomic medicine. Other clinical information of the type collected by treating physicians and stored in electronic medical records will also be collected to aid in the interpretation of laboratory data. Participants will also be asked to consent for future access of the medical record, future research on biospecimens and data generated from genomic sequencing, and for the ability to re-contact.

As part of this effort, Nicklaus Children's Hospital plans to create a large integrated database that contains the DNA sequences of the participants' whole human genomes and additional health information regarding characteristics and health of the persons whose samples have been sequenced. Scientists can then use the database to try to link those traits, diseases, and other conditions to changes in the sequence of the genome. Nicklaus Children's Hospital plans to make the database available to its collaborators, such as RCIGM, pharmaceutical and biotechnology companies, and other academic institutions which will use the database to find better, innovative ways to prevent, diagnose, and treat cancer and other diseases. De-identified data from this study will be shared with the community at-large, including publications and public databases. In addition, participants will be given the option to allow biospecimens (i.e., residual blood, saliva, CSF, etc.) to be included in biorepositories at Nicklaus Children's Hospital and Rady Pediatric Genomics & Systems Medicine Institute (RCIGM).

The study will provide clinical laboratory-confirmed results related to the affected patient's phenotype, including optional incidental findings unless subjects opt-out for these additional results, to allow for these research findings to be used in clinical care. Furthermore, this study will aggregate data regarding standard clinical genetic testing as well as cost measures to not only identify differences in diagnostic rates, diagnostic accuracy, and times to diagnoses, but to determine the cost-effectiveness of this testing and subsequent changes in care management. Clinical utility will be defined as changes in care that follow directly from results of genetic testing (both positive and negative), including standard clinical tests and WGS. This data will be used to further examine the analytic, diagnostic, and clinical utility and cost-effectiveness of this testing.

WGS methods continue to improve and pediatric genomic medicine is a very new field of medical practice. This study will also inform investigators regarding best practices, both in terms of traditional medical outcomes and patient-centered outcomes. Consequently, this study will also act as a biorepository for samples and data as the ability to share genomic and phenotypic data amongst researchers is critical to progressing our understanding of the nascent field of pediatric genomic medicine.

Specific Aims:

1. Use WGS to identify new genetic diagnoses in children with multiple congenital anomalies, developmental delay, autism, seizures, intellectual disabilities, neurodegenerative disorders, and metabolic illness.
2. Evaluate the diagnosis rate of genetic diseases by WGS in previously undiagnosed patients.
3. Assess the clinical utility of WGS in the care and management of patients.
4. Examine the health economics and cost-effectiveness of WGS.
5. Evaluate the provider, patient and family experience with genomic medicine
6. Collect biological samples and associated clinical data from pediatric patients who may have a genetic disease and their family members (the "Phenome").
7. Create, analyze and store genomic data from the biological samples. Genomic data will include genomic (gDNA) sequences, RNA sequences, and/or other related 'omic data (including, but not limited to, pharmacogenomics, transcriptomics, and epigenomics). Genomic data from WGS will include single nucleotide variants (SNVs), structural variants such as copy number testing, genomic rearrangements, gene expression , the "whole transcriptome" or more limited DNA sequencing panels of specific genes or of all exons of genes (the "Exome").
8. Analyze and report clinically-confirmed genomic diagnoses and treatment guidance through use of new research technologies.
9. Identify and study novel gene and disease processes.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic male or female children ages 0-21 who have un unknown medical condition thought to have an underlying genetic cause after parental consent has been obtained.
* Willingness of referring provider or other qualified medical staff member to participate in this study by facilitating collection of biologic specimens and clinical information.
* Patient whose medical condition can be reasonably attributed to a possible genetic etiology.
* Patient have had at least one diagnostic test without a definite diagnosis.

Exclusion Criteria:

* Unwillingness to consent to research.
* Affected adults (>21 years of age), unless they are a biological relative of the affected child.
* Any patient whose medical condition cannot be reasonably attributed to a possible genetic etiology or there is a prior diagnosis that explains the child's clinical presentation.

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children from 0 to 21 years suffering from unknown diagnoses seen at Nicklaus Children's Hospital
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2018-02-20 (Actual); Primary Completion 2070-03 (Estimated); Study Completion 2070-03 (Estimated)

PRIMARY OUTCOMES:
Number of patients enrolled per year | Yearly throughout study completion up to 50 years
  Total number of enrolled patients who will undergo WGS testing

SECONDARY OUTCOMES:
Diagnosis Rate of genetic diseases | Throughout study completion up to 50 years
  Proportion of diagnosis rate of genetic diseases by WGS in previously undiagnosed patients
Clinical Utility | Throughout study completion up to 50 years
  Total number of clinical utility of WGS in the case and management of patients
Phenome | Throughout study completion up to 50 years
  Total number of biological samples and associated clinical data who have a genetic disease and their family members
Clinically-confirmed diagnoses | Throughout study completion up to 50 years
  Proportion of clinically-confirmed genomic diagnoses and treatment guidance through the use of new research technologies

CONTACTS AND LOCATIONS:
Overall Officials: Parul Jayakar, MD, Principal Investigator — Nicklaus Children's Hospital
Locations (1):
- Nickalus Children's Hospital f/k/a Miami Children's Hospital, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] McCandless SE, Brunger JW, Cassidy SB. The burden of genetic disease on inpatient care in a children's hospital. Am J Hum Genet. 2004 Jan;74(1):121-7. doi: 10.1086/381053. Epub 2003 Dec 12. PMID 14681831
- [Background] Sawyer SL, Hartley T, Dyment DA, Beaulieu CL, Schwartzentruber J, Smith A, Bedford HM, Bernard G, Bernier FP, Brais B, Bulman DE, Warman Chardon J, Chitayat D, Deladoey J, Fernandez BA, Frosk P, Geraghty MT, Gerull B, Gibson W, Gow RM, Graham GE, Green JS, Heon E, Horvath G, Innes AM, Jabado N, Kim RH, Koenekoop RK, Khan A, Lehmann OJ, Mendoza-Londono R, Michaud JL, Nikkel SM, Penney LS, Polychronakos C, Richer J, Rouleau GA, Samuels ME, Siu VM, Suchowersky O, Tarnopolsky MA, Yoon G, Zahir FR; FORGE Canada Consortium; Care4Rare Canada Consortium; Majewski J, Boycott KM. Utility of whole-exome sequencing for those near the end of the diagnostic odyssey: time to address gaps in care. Clin Genet. 2016 Mar;89(3):275-84. doi: 10.1111/cge.12654. Epub 2015 Sep 22. PMID 26283276